CLINICAL TRIAL: NCT06355362
Title: Association of Intraoperative Hemodynamic Characteristics to Postoperative Complications and Mortality
Acronym: HeCoMo
Status: Not yet recruiting | Type: Observational
Sponsor: Kliniken Essen-Mitte (Other)
Responsible Party: Sponsor
Other Study IDs: HeCoMo
Record Dates: First submitted 2024-03-19; First posted 2024-04-09 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: High-risk Surgery
Keywords: hemodynamic; transfusion; perioperative process quality; intensive care medicine; complications; mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Worldwide, about 400 million major surgeries are performed annually. The scarce data available in the literature still suggest high postoperative morbidity and mortality, even in Europe. Data of the World Health Organization on causes of death suggest that death after surgery would be the number three cause of mortality if it were considered a separate cause of death. However, there is little structured or high-quality data on postoperative mortality in the literature.

The aim of this study project is to collect data on postoperative complications and mortalities worldwide and to establish a Perioperative Outcome Study Platform on this topic.

In the first study of this platform, we aim to investigate the association of hemodynamic characteristics with postoperative complications and mortality. It is a prospective, multi-center study.

In addition, the investigators aim to collect data on the structural characteristics of the study sites and, for each patient, characteristics of quality of perioperative care in order to analyze associations with hemodynamic characteristics and postoperative complications and mortalities.

DETAILED DESCRIPTION:
Preamble

The Perioperative Outcome (POP-OUT) project aims to improve care for our patients and intends to build a community of physicians from all over the world being dedicated to that aim.

The purpose and vision of the Perioperative Outcome study project

In perioperative care outcome data about postoperative mortality and morbidity is rare. This project aims to fill that gap with a prospective international database collecting perioperative data of surgical patients and relate them to postoperative mortality and morbidity.

The project is planned as initial observational study to build up the structures and define the case. Subsequently, based on that initial project the investigators further develop the study platform. This platform should adapt, grow, and broaden according to the results and possibilities seen in the study generations year by year. The intention is not to set-up a study group that finishes its work if the study is performed, but they hand on the study to the next generation of the community.

The vision is that in the future the outcome data offer the possibility to diversify, plan and power statistically prospective intervention trials to address the mortality and morbidity of our patients.

The idea is to establish a global community of anesthetists and intensivists to develop such a study platform together. The community is stronger than everything else.

The first steps of the study platform

The goal is to start with an initial observational trial about hemodynamic perioperative characteristics (fluids, vasopressors, inotropes, transfusions, hypotensive events) and short- and long-term outcomes.

The outcome measures should be in the short-term postoperative complications according to the classification of CLAVIEN-DINDO greater or equal to IIIb (example lists will be provided to the community, but the main point is that greater or equal to the category IIIB requires an intervention making it transparent in the documentation process).

The long-term outcome will be mortality (in-hospital, three-months, or one-year mortality).

The working title should be: "Association of Hemodynamic characteristics to postoperative Complications and Mortality" with the short title: "HeCoMo".

But it is like a pilot trial offering us the possibility to build up a platform structure to continuously develop perioperative outcome studies in all fields of perioperative care.

Which patients to include in the first observational trial

The initial main study population will be high-risk surgery, but this is not limited nor fixed for now nor for future projects.

It will be up to the community which specialties we will include or if we stratify the surgical populations, but the actual plan is to define a positive list of surgeries to be included. As example we can list for abdominal procedures:

* esophageal resection
* gastric resection with intestinal anastomosis
* pancreatic resections (whole organ, head, or tail)
* multivisceral procedures, e.g., cancer debulking due to ovarian cancer
* urological cystectomies.

Study aims of the initial observational trial

The primary hypothesis of the first observational trial is to test which hemodynamic measures are associated to postoperative morbidity or mortality. The measures to test are the cumulative amount and the longitudinal aspects of the intraoperative values of:

* intravenous infusion volume
* fluid balance
* hypotensive events
* vasopressor administration
* administration of inotropes
* any type of transfusions

It must be stated that the innovation of the study is not the study design nor its fancy primary outcome measures or statistical analysis. The issue is that it is a question not explicitly addressed in the literature and international short- and long-term outcome are not available in this context.

The idea is that every center includes 15-25 patients in the sequence of their appearance.

But nevertheless, the study goal is of clinical relevance and will offer the opportunity to be published at a good scientific level.

Data management

An important feature is that the data should belong to the community. That means that after the initial primary publication of every study generation the data can be used for subsequent sub-analysis or to plan subsequent powered intervention studies. At the end the long-term goal of that project is that the data are owned by the community.

The development of the electronic case report form is planned. The data acquisition will be in RedCap hosted on the server and the management of the Evangelische Kliniken Essen-Mitte, Essen, Germany by the Department of Anesthesiology, Intensive Care Medicine, and Pain therapy.

The data can be entered in the system via a webpage or via smartphone or tablet online and offline.

Ethical consent and vote by the competent authority

Obtaining an ethical vote by the competent authority and depending on the vote perceiving informed consent is up to the local institutions. In some countries it may be possible to conceive a waiver of individual patient consent. But this must be cleared out at the national level by the national coordinators. An important argument for the waiver is that the study population is more representative and is not biased by selection bias. Additionally, the study participation is expected at no additional risk for the study patients.

The general idea is that this project is a prospective, indefinite database related to perioperative outcome with sub-questions regarding hemodynamic, respiratory, metabolic, etc. issues.

Funding of the project

It is important to state that this project will have no funding by a medical society or any other entity. To be independently the study should be based by the voluntary activities of their contributors or by the departmental funding of any involved institution. However, during the development of the study platform it can be required to receive funding for maintaining data management structures or similar requirements. If the steering committee agrees on such a particular funding approach the community will be informed.

The structure of the study group

The idea is to define a steering committee and national coordinators. They are granted co-authorship for the resulting publication. But everybody taking responsibility and care of the project will be mentioned in the acknowledgements.

An exact statement about authorship of any analysis of the project will be send to everybody involved in the study platform prior to the inclusion of the first study patient.

The national coordinators take responsibility of the organization and recruitment of the study centers within his/her own country or region.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgery with increased postoperative morbidity and/or increased postoperative mortality

Exclusion Criteria:

* Patients undergoing surgery in the field of obstetrics
* Age < 18 years
* Lack of written informed consent
* Lack of language understanding
* Unwillingness to store disease data on site and share anonymised data as part of the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The decision as to whether a surgical procedure has an increased risk of postoperative complications and/or postoperative mortality is the responsibility of the study leader at the respective study site. The list of surgical procedures will be agreed between the study site and the head of the study. The presence or absence of co-morbidities is not included in the assessment of perioperative risk.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative complications | From the time of surgery up to hospital discharge or up to the 30th postoperative day
  The postoperative complications are graded according to the CLAVIEN-DINDO classification
Incidence of postoperative mortalities | From the time of surgery up to one year after surgery, during hospital stay, at three, six, or twelve months after surgery
  The incidence of postoperative mortality during the follow-up period

SECONDARY OUTCOMES:
Implementation rate of preoperative factors impacting postoperative outcome | During the 48 hours prior to surgery
  Implementation rate in percentage of preoperative factors like fasting periods, preoperative carbohydrate drinks or the use of bowel preparations
Intraoperative hemodynamic characteristics | Time period during surgery
  The longitudinal course and punctual values during surgery of haemodynamic parameters like heart rate and mean arterial pressures and therapies such as infusion volumes and balances, and catecholamine administration
Postoperative haemodynamic characteristics | Time period from the end of surgery up to the third postoperative day
  The longitudinal course and punctual values after surgery up to the third postoperative day of haemodynamic parameters like heart rate and mean arterial pressures and therapies such as infusion volumes and balances, and catecholamine administration
Co-morbidities of patients | At the day of surgery
  Descriptive data about the co-morbidities of the study patients
Transfusion of blood components and administration of coagulation factors | During hospital stay or up to the 30th postoperative day
  The number of transfusions of packed red blood cells, plasma, or thrombocytes as well as coagulation factors per patients
Score of the physical/pathological activity status of the patients | During the 48 hours prior to surgery
  Score of the the exercise ability in metabolic equivalent of task units
Clinical frailty scale | During the 48 hours prior to surgery
  Score according to the clinical frailty scale in categories 1 to 9
Characteristics of perioperative care, time in perioperative units and the hospital | During hospital stay or up to the 30th postoperative day
  Length of patient stay in the hospital, time pre- and postoperatively in hospital, stay in recovery room, post-anesthesia care unit, intensive care medicine.
Characteristics of provision of anesthesia and type of pain therapy | Time period from the start of anaesthesia up to the third postoperative day
  Data about the type of anaesthesia and the drugs used with their doses as well as the drugs and methods and drugs to control pain
Implementation rate of items perioperatively impacting outcome within an Enhanced-Recovery-After-Surgery pathway description | During hospital stay or up to the 30th postoperative day
  The implementation rate in percentage of perioperative items related to perioperative treatment modalities

CONTACTS AND LOCATIONS:
Overall Officials: Aarne Feldheiser, Principal Investigator — Kliniken Essen-Mitte

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Webpage of the study platform — https://www.popoutstudy.org/index.html